CLINICAL TRIAL: NCT02848300
Title: Evaluation of Local Pharmacokinetics and Tolerability of Bimatoprost Applied Topically to the Scalp of Male Patients With Androgenetic Alopecia
Brief Title: Local Pharmacokinetics and Tolerability of Bimatoprost Applied to the Scalp of Male Patients With Androgenetic Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1666-101-012
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Bimatoprost 1% Formulation A solution applied to the left side of the scalp and trunk area and Bimatoprost 1% Formulation B solution applied to the right side of the scalp and trunk area once daily for 14 days.
  Interventions: Drug: Bimatoprost 1% Formulation A; Drug: Bimatoprost 1% Formulation B

INTERVENTIONS:
Drug: Bimatoprost 1% Formulation A — Bimatoprost 1% Formulation A solution applied to the scalp and trunk once daily for 14 days.
Drug: Bimatoprost 1% Formulation B — Bimatoprost 1% Formulation B solution applied to the scalp and trunk once daily for 14 days.

SUMMARY:
This study will evaluate the skin pharmacokinetics and tolerability of bimatoprost Formulation A and Formulation B following 14 days of once daily topical administration in male participants with androgenetic alopecia (AGA).

DETAILED DESCRIPTION:
Single-center, multiple-dose study evaluting the local pharmacokinetics and tolerability of bimatoprost following 14 days of once daily topical administration of bimatoprost Formulation A and Formulation B (both containing 1% bimatoprost) to the scalp of male patients With androgenetic alopecia

ELIGIBILITY:
Inclusion Criteria:

-Patients with mild to moderate Androgenetic Alopecia of the vertex area of the scalp.

Exclusion Criteria:

* Patients with uncontrolled systemic disease
* History of significant cardiovascular disease
* Scarring disease, infection, or abnormality of the scalp or hair shaft or systemic disease that could cause temporary hair loss (eg, seborrheic dermatitis, psoriatic dermatitis, alopecia areata, cicatricial alopecia, uncontrolled hyperthyroidism/hypothyroidism, tinea infections, and genetic disorders)
* Patients who have received hair transplants or have had scalp reductions
* Abnormal bone biomarker laboratory results.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Drug Concentration in Skin Biopsy Samples | Day 14
Percentage of Participants with at Least 1 Treatment Emergent Adverse Event | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Danielle McGeeney, Study Director — Allergan
Locations (1):
- DermResearch, LLC, Austin, Texas, United States